CLINICAL TRIAL: NCT05152706
Title: Parkinson´s Disease, Aerobic Exercise and Photobiomodulation: a Randomised Controlled Trial
Brief Title: Parkinson´s Disease, Aerobic Exercise and Photobiomodulation
Acronym: PDAERPBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Luis Santos, Principal Investigator, University of Oviedo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: No. 295/19
Record Dates: First submitted 2021-11-28; First posted 2021-12-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention aerobic (IAER) (Experimental): Patients assigned to the IAER participated in fourty-eigth aerobic exercise therapy sessions over the course of six months.
  Interventions: Other: Aerobic training
- Intervention photobiomodulation (IPBM) (Experimental): Patients assigned to the IPBM participated in fourty-eigth transcraneal photobiomodulation (PBM) theraphy sessions, using a therapeutic laser console, over the course of six months.
  Interventions: Other: Photobiomodulation
- Intervention aerobic and photobiomodulation (IAER+PBM9 (Experimental): Patients assigned to the IAER+PBM participated in the aerobic exercise therapy and the PBM one at the same time, during six months.
  Interventions: Other: Aerobic training; Other: Photobiomodulation
- Control (CO) (No Intervention): Patients assigned to the control (CO) did not participated in any kind of therapy, they just followed their usual weekly routine during six months

INTERVENTIONS:
Other: Aerobic training — Cycling at the aerobic intensity
  Arms: Intervention aerobic (IAER); Intervention aerobic and photobiomodulation (IAER+PBM9
Other: Photobiomodulation — Photons therapy
  Arms: Intervention aerobic and photobiomodulation (IAER+PBM9; Intervention photobiomodulation (IPBM)

SUMMARY:
The aim of the present study was to assess the effects of a combined therapy of aerobic exercise and transcranial photobiomodulation upon the cardinal motor sympomts of Parkinson´s disease of a group of Parkinson´s disease patients. It was hypothesized that aerobic exercise and transcranial photobiomodulation would yield significant benefits in the cardinal motor sympomts of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with idiopathic PD and rated 1-2 on the Hoehn and Yahr Scale.
* No type of dementia as assessed by the mini-mental state examination.
* Able to stand for 2 min without assistance.
* Able to walk 10 m without assistance.

Exclusion Criteria:

* Individuals were excluded if they suffered a neurological disease other than PD, if the subject has an implant of any kind in the head (e.g., stent, clipped aneurysm, embolized arteriovenous malformation, implantable shunt - Hakim valve) or if they did not meet the eligibility criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
MDS-UPDRS | 6 months
  The motor portion of the Movement Disorder Society-Unified Parkinson´s (MDS-UPDRS, the minimum and maximum values are 0 and 72, respectively and the higher score, the worse patient condition)

SECONDARY OUTCOMES:
DASH | 6 months
  The disabilities of the arm, shoulder and hand (DASH, the minimun and maximum values are 0 and 190, respectively and the higher score, the worse patient condition)
Static posturography | 6 months
  The centre of pressure (CoP) parameters (these CoP parameters; Length, in mm, Area in mm2 and Speed, Xspeed and Yspeed in m/s will be combined to report the static posturography)
TMWT | 6 months
  10 meters walking test (speed in seconds)
TUG | 6 months
  Time up Go Test (speed in seconds)
Grip strength | 6 months
  Grip strength in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education and Sport, University of León, León, Castille and León, Spain

REFERENCES:
- [Derived] Santos L, Burtscher J, de Taboada L. Parkinson's disease, aerobic exercise and photobiomodulation: a randomised controlled trial. J Neural Transm (Vienna). 2025 Oct 31. doi: 10.1007/s00702-025-03050-7. Online ahead of print. PMID 41171380